CLINICAL TRIAL: NCT04561401
Title: Can Brain Stimulation Enhance Outcomes Associated With Intensive Rehabilitation for Youth With Chronic Pain?
Brief Title: IPRP Repeated Transcranial Magnetic Stimulation (rTMS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Jillian Vinall Miller, Assistant Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB20-1464
Record Dates: First submitted 2020-09-11; First posted 2020-09-23 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- rTMS + IPRP (Experimental): 25 youth aged 10-18 years with severe chronic pain will be invited to partake in the Intensive Pain Rehabilitation Program, where they will receive Repeated Transcranial Magnetic Stimulation as one of their treatment interventions.
  Interventions: Device: Repeated Transcranial Magnetic Stimulation (rTMS); Other: Intensive Pain Rehabilitation Program (IPRP)
- IPRP (Active Comparator): Youth within this arm will not be receiving the rTMS intervention. Rather, they will only be enrolled within the IPRP.
  Interventions: Other: Intensive Pain Rehabilitation Program (IPRP)

INTERVENTIONS:
Device: Repeated Transcranial Magnetic Stimulation (rTMS) — rTMS will be applied at 10 Hz. Each train will consist of 40 supra threshold (120% resting motor threshold) pulses over 4 seconds with an inter-train interval of 26 seconds. Treatment sessions will last 37.5 minutes (75 trains/3,000 pulses), and occur at the same time of day on every weekday for a period of three weeks (15 days total). During TMS, only passive activities will be allowed (i.e., watching movies or TV, listening to music). Three weeks of treatment was selected based on existing rTMS evidence in youth with treatment resistant major depressive disorder.
  Arms: rTMS + IPRP
Other: Intensive Pain Rehabilitation Program (IPRP) — The paediatric Intensive Pain Rehabilitation Program (IPRP) in Canada was established to target youth with severe chronic pain and consequent functional disability who do not respond to standard outpatient pain therapies. The IPRP at the Alberta Children's Hospital (ACH) involves three- to six-weeks of day-treatment rehabilitation, provided by an interdisciplinary team (e.g. Psychology, Physiotherapy, Family Therapy). This rehabilitative program teaches self-management strategies with the goal of helping youth and their families resume normal daily functioning.

SUMMARY:
Severe chronic pain is defined as pain persisting for three months or more that significantly impacts daily functioning. It is highly prevalent, occurring in 100,000 to 160,000 youth. If left unmanaged it can lead to persistent pain and mental health problems in adulthood, posing enormous costs to society ($7.2 billion CAD/year). In 2014, health professionals at the Alberta Children's Hospital (ACH) established a pediatric Intensive Pain Rehabilitation Program (IPRP) to target youth with severe chronic pain and consequent functional disability who do not respond to outpatient pain therapies. The IPRP at the ACH is a three-week intensive day-treatment intervention provided by an interdisciplinary team, which helps youth resume engagement in normal daily functioning. Following IPRP, youth reported less anxiety, less depressive symptoms, and greater function, although their self-reported pain remained unchanged. In August 2016, the investigators began to explore brain areas related to severe chronic pain in youth. The investigators scanned a subset of youth at the start (baseline) and end (discharge) of IPRP (23 youth with 2 brain scans). From baseline to discharge, the investigators saw decreases in activity in the dorsolateral prefrontal cortex (DLPFC). Decrease in DLPFC activity was related to better mental health outcomes. The DLPFC is a well-known target for non-invasive brain stimulation. Repeated brain stimulation has been used to treat adults, but not youth with chronic pain. For the first time, the investigators will use image-guided brain stimulation (37 minutes/day, 5 days/week) to enhance the brain changes observed with IPRP. The investigators will examine whether three weeks of brain stimulation helps to reduce pain symptoms in youth. The investigators will also compare pain, brain, and mental health outcomes to our historical program data. By adding brain stimulation to our pain intervention, the investigators have the chance to target an area of the brain investigators know to be altered by chronic pain to improve outcomes.

DETAILED DESCRIPTION:
Severe chronic pain in youth is debilitating, common, and has limited treatment options, rendering it as a major public health problem. Severe chronic pain is defined as pain persisting for three months or more that significantly impacts daily functioning (e.g. sleep, mental health, school, work, activity). It is highly prevalent, occurring in 100,000 to 160,000 youth in Canada - comparable to the rates of autism spectrum disorder. If left unmanaged, it can lead to persistent pain and mental health problems in adulthood, posing enormous costs to society ($7.2 billion CAD/year). Most treatments to address chronic pain take a "one-size-fits-all-approach," which does not account for comorbid mental health conditions, contributing to small treatment effects.

In 2014, the Vi Riddell Children's Pain and Rehabilitation Program at the Alberta Children's Hospital (ACH) established the first pediatric Intensive Pain Rehabilitation Program (IPRP) in Canada to target youth with severe chronic pain and consequent functional disability who do not respond to standard outpatient pain therapies. The IPRP at the ACH involves three- to sex-weeks of day-treatment rehabilitation, provided by an interdisciplinary team (e.g. Psychology, Physiotherapy, Family Therapy). This rehabilitative program teaches self-management strategies with the goal of helping youth and their families resume normal daily functioning. Similar to other intensive rehabilitation programs, at discharge from IPRP, youth reported less anxiety, less depressive symptoms and better functioning, although, their self-reported pain intensity remained unchanged. It is generally thought that by returning to normal daily activities, youth will learn to function with their pain, and their pain will dissipate over time. However, there is limited evidence to support this. Long-term follow-up of youth in IPRP revealed a reduction of pain interference in daily activities. However, at one-year post-IPRP, youth's self-reported ratings of depression and quality of life did not differ from their ratings prior to completing IPRP. In order to improve long-term recovery and reduce the burden of suffering on the individual, their family and society, evidence-based and targeted interventions are needed to reduce pain and pain-related disability in youth with severe chronic pain.

For a chronic pain treatment to be evidence-based, it needs to draw on the known neurobiological and psychological processes underlying the development and maintenance of severe chronic pain. In August 2016, investigators began scanning a subset of youth in our IPRP at baseline and again at discharge from the program. Preliminary analysis of this neuroimaging data (23 youth with 2 scans each) suggested decreased functional responses to emotional stimuli in the dorsolateral prefrontal cortex (DLPFC) from baseline to discharge of affected youth, commensurate with decreases in internalizing mental health symptoms.

The DLPFC is a large and functionally heterogeneous brain region. It is generally associated with driving appropriate behavioral responses, and top-down modulation. Therefore, with regards to pain it has been shown to be involved in both pain detection and in pain suppression. Given its involvement in pain modulation, it is feasible that the DLPFC could serve as a therapeutic target.

By targeting the DLPFC using repetitive transcranial stimulation (rTMS), the investigators may be able to enhance outcomes associated with IPRP. Work from our institution demonstrated that rTMS of the DLPFC is a safe and effective method for treating youth with treatment resistant major depressive disorder. In addition to treatment resistant major depressive disorder, rTMS of the DLPFC has also been found to be effective in managing chronic pain in adults. rTMS uses a magnetic field to non-invasively stimulate small targeted regions of the brain. The magnetic coil produces small electric currents in the region of the brain just under the coil via electromagnetic induction. Magnetic resonance imaging (MRI) can be used to help identify and target specific brain regions, such as the DLPFC, providing an individualized approach to treat the patient's symptoms. To date, rTMS has not been utilized to manage pain and comorbid mental health conditions in youth. Using an open-label clinical trial study design, the investigators will examine whether the addition of rTMS to IPRP reduces pain intensity and enhances brain and behavioral changes associated with standard IPRP care to improve outcomes of youth with severe chronic pain.

Aim 1: Determine whether rTMS in addition to IPRP reduces self-reported pain intensity from baseline to discharge in youth with severe chronic pain. Hypothesis 1: The addition of rTMS to IPRP will result in decreases in self-reported pain intensity from baseline to discharge in youth with severe chronic pain.

Aim 2: Examine whether youth that undergo rTMS in addition to IPRP versus IPRP alone have greater improvements in outcomes from baseline to discharge. Hypothesis 2: The addition of rTMS to IPRP will result in greater decreases in DLPFC responsivity to emotional stimuli and greater decreases in self-reported pain intensity, functional disability, anxiety, depressive and post traumatic stress disorder (PTSD) symptoms between baseline and discharge as compared to youth that underwent the standard IPRP.

Aim 3: Examine whether changes following IPRP persist beyond discharge in youth that underwent rTMS in addition to IPRP versus IPRP alone. Hypothesis 3: Parent and self-reported.

Methods: Between November 2020-2023, 25 youth aged 10-18 years with severe chronic pain will be invited to partake in IPRP. In addition to the standard three-week IPRP, youth will receive an rTMS intervention utilizing a robot-controlled, Magstim SuperRapid2, air-cooled 90mm figure-of-8-coil (Magstim, Wales UK). Following standardized protocols for youth with treatment resistant major depressive disorder, rTMS will be applied to the individual's DLPFC as defined by functional imaging for 37.5 minutes per weekday, at the same time of day, for a period of three weeks (15 days total). Participants will be monitored for adverse events and tolerability using a Pediatric TMS Safety and Tolerability Measure (20) on days 1, 6, and 11. Youth will undergo a 3T MRI at baseline and discharge from IPRP. Both structural and functional images will be acquired. At baseline and discharge, youth will also complete a battery of reliable and validated questionnaires assessing pain, functional disability, anxiety, depressive and PTSD symptoms.

rTMS: Motor evoked potentials will be recorded to determine the resting motor threshold. Initially, to locate the DLPFC target site, the five centimetre rule will be applied in which the scalp position five centimetres anterior to the hotspot along a line to the nation will be marked. Using a neuronavigation system (Brainsight2, Rogue Research, Montreal), the TMS coil will be monitored in real time and co-registered with the individual's functional MRI. Neuronavigation will be used to confirm accurate DLPFC targeting. The TMS coil will subsequently be placed tangential to the scalp, and angled at 45 degrees to the midline and fixed over the DLPFC using a mechanical arm.

rTMS will be applied at 10 Hz. Each train will consist of 40 threshold (100% resting motor threshold) pulses over 4 seconds with an inter-train interval of 26 seconds. Treatment sessions will last 37.5 minutes (75 trains/3,000 pulses), and occur at the same time of day on every weekday for a period of three weeks (15 days total). During TMS, only passive activities will be allowed (i.e., watching movies or TV, listening to music). Three weeks of treatment was selected based on existing rTMS evidence in youth with treatment resistant major depressive disorder.

Neuroimaging: Cortical volumes will be acquired from a T1-weighted anatomical scan. FreeSurfer will be used for processing, editing, and segmenting structural brain images. The automated recon-all pipeline will be used to perform brain extraction, image registration, motion and intensity correction, and segmentation/parcellation. Each image will be manually checked, and cortical volumes will be extracted.

Functional magnetic resonance imagine (fMRI) will be used to detect blood oxygen level-dependent (BOLD) signal changes during the presentation of validated pictures of facial affect that were used in the previous IPRP neuroimaging study. This paradigm consists of 36, standardized photos from female and male individuals depicting neutral, happy and fearful facial expressions. These photos will be randomized into 4 blocks presented 4 times, and each face will be presented for 200-ms with a 300-ms interstimulus. The investigators will apply standard preprocessing (slice-time correction, B0-unwarping, motion correction, bandpass temporal filtering, template registration and smoothing) in SPM. Motion will be censored using the ART toolbox. Second-level analyses will be used to compare differences in contrasts over time and between groups. All statistical tests will be corrected for multiple comparisons (cluster-corrected false discovery rate q<0.05, with cluster-forming height threshold of p<0.001).

Finally, a resting-state fMRI scan will be acquired and undergo standard preprocessing in SPM. Motion will be censored using the ART toolbox. Cortical masks derived from FreeSurfer will be used as seed regions for fMRI functional connectivity analysis. Time courses for the DLPFC will be extracted and used as a regressor to identify correlations with all other brain regions. Second-level analyses will be used to test differences in functional connectivity over time and between groups. All statistical tests will be corrected for multiple comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 10-18 years
* Patient has had the appropriate medical work-up
* Participation in accessible, evidenced based pain therapies has not demonstrated return to functional goals
* Pain is significantly impacting the patient's life and they are not meeting their functional goals in areas of life, which may include: physical function, sleep, self-care, school attendance/academic performance, social function, recreational engagement, and mood
* Patient and family agree and understand that an active, self-management approach to functional restoration is the mainstay of treatment in the IPRP

Exclusion Criteria:

* Significant developmental delay or brain injury
* Functional neurological disorder/conversion disorder
* Youth who require opioid weaning
* Extensive medical needs and/or untreated psychiatric illness that would impede a rehabilitative approach to care.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-10-19 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Pain Presence | This outcome will be measured at baseline.
  The commonly used Pain Questionnaire will be administered to measure the presence and characteristics of pain. Youth will rate the average frequency ("not at all" to "daily"), duration ("less than 1 hour" to "all day"), and intensity ("no pain" to "worst pain possible") of their pain.
Pain Frequency | This outcome will be measured at baseline.
  The commonly used Pain Questionnaire will be administered to measure the presence and characteristics of pain. Youth will rate the average frequency ("not at all" to "daily"), duration ("less than 1 hour" to "all day"), and intensity ("no pain" to "worst pain possible") of their pain.
Pain Duration | This outcome will be measured at baseline.
  The commonly used Pain Questionnaire will be administered to measure the presence and characteristics of pain. Youth will rate the average frequency ("not at all" to "daily"), duration ("less than 1 hour" to "all day"), and intensity ("no pain" to "worst pain possible") of their pain.
Pain Intensity | This outcome will be measured at baseline.
  The commonly used Pain Questionnaire will be administered to measure the presence and characteristics of pain. Youth will rate the average frequency ("not at all" to "daily"), duration ("less than 1 hour" to "all day"), and intensity ("no pain" to "worst pain possible") of their pain.
Pain Interference | This outcome will be measured at baseline.
  Youth will complete the Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Profile-25. The Pain Interference subscale uses 4 items to assess whether pain has interfered with youth's everyday activities in the past 7 days using a 5-point Likert scale (anchors: 0 = "never" and 4 = "almost always"). The PROMIS measures demonstrated good construct validity (intercept and slope equal or greater to 0.98) and internal consistency (pain interference, 4 items alpha = 0.85).
Brain imaging | This outcome will be measured at baseline (upon admittance into the program).
  Structural and functional imaging will be acquired using resting-state functional magnetic resonance imaging (fMRI) scan. Motion will be censored using the Artifact Detection Tools (ART). Cortical masks derived from FreeSurfer will be used as seed regions for fMRI functional connectivity analysis. Time courses for the dorsolateral prefrontal cortex (DLPFC) will be extracted and used as a regressor to identify correlations with all other brain regions. Second-level analyses will be used to test differences in functional connectivity over time and between groups. All statistical tests will be corrected for multiple comparisons.
Functional disability | This outcome will be measured at baseline.
  The Functional Disability Inventory (FDI) will be administered to assess functional disability. Youth will rate their level of difficulty in completing daily activities in a variety of settings (e.g. home, school) on a 5-point Likert scale ranging from 0 "no trouble" to 4 "impossible." Higher scores are indicative of greater pain-related disability. The FDI has high internal consistency at baseline (alpha = .90) and post-treatment (alpha = .87).
Anxiety and Depressive Symptoms | This outcome will be measured at baseline.
  Anxiety and depressive symptoms will be assessed using the PROMIS Pediatric Profile-25 Anxiety and Depression subscales. Participants will report if they experienced any of the symptoms in the past 7 days using a 5-point Likert scale (anchors: 0 = "never" and 4 = "almost always"). The subscales have demonstrated good construct validity (intercept and slope equal to or greater than 0.93) and excellent internal consistency (depressive symptoms, 4 items, alpha = 0.91; anxiety symptoms, 4 items, alpha = 0.90).
Posttraumatic Stress Disorder (PTSD) Symptoms | This outcome will be measured at baseline.
  Youth PTSD symptomology will be assessed using the Child PTSD Symptom Scale (CPSS-V). The CPSS-V is a 20-item measure that maps on to the Diagnostic and Statistical Manual of Mental Disorders 5th Edition PTSD criteria, and assessed PTSD symptoms experienced by youth in the past month. Youth will be asked to identify something scary or upsetting that bothers them to think about. With that event in mind, they will be asked to respond to 20 items assessing PTSD symptoms on a 5-point Likert scale, ranging from "not at all" to "6 or more times a week/almost always." Total symptom severity scores are obtained by summing the 20 items (range: 0-80). A score of 31 or above indicates clinically elevated PTSD symptoms. The CPSS-V has excellent internal consistency, good test-retest reliability, and good convergent validity.
Pediatric Transcranial Magnetic Stimulation (TMS) Safety and Tolerability | This outcome will be measured at Day 1.
  Possible adverse events (headache, presyncope, nausea, etc.) will be screened and quantified as either mild, moderate, or severe. Any other potential side effects will be recorded and quantified.
Pain Presence | This outcome will be measured at discharge from the program, which is approximately 3 weeks from the time of admittance.
  The commonly used Pain Questionnaire will be administered to measure the presence and characteristics of pain. Youth will rate the average frequency ("not at all" to "daily"), duration ("less than 1 hour" to "all day"), and intensity ("no pain" to "worst pain possible") of their pain.
Pain Frequency | This outcome will be measured at discharge from the program, which is approximately 3 weeks from the time of admittance.
  The commonly used Pain Questionnaire will be administered to measure the presence and characteristics of pain. Youth will rate the average frequency ("not at all" to "daily"), duration ("less than 1 hour" to "all day"), and intensity ("no pain" to "worst pain possible") of their pain.
Pain Duration | This outcome will be measured at discharge from the program, which is approximately 3 weeks from the time of admittance.
  The commonly used Pain Questionnaire will be administered to measure the presence and characteristics of pain. Youth will rate the average frequency ("not at all" to "daily"), duration ("less than 1 hour" to "all day"), and intensity ("no pain" to "worst pain possible") of their pain.
Pain Intensity | This outcome will be measured at discharge from the program, which is approximately 3 weeks from the time of admittance.
  The commonly used Pain Questionnaire will be administered to measure the presence and characteristics of pain. Youth will rate the average frequency ("not at all" to "daily"), duration ("less than 1 hour" to "all day"), and intensity ("no pain" to "worst pain possible") of their pain.
Pain Interference | This outcome will be measured at discharge from the program, which is approximately 3 weeks from the time of admittance.
  Youth will complete the Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Profile-25. The Pain Interference subscale uses 4 items to assess whether pain has interfered with youth's everyday activities in the past 7 days using a 5-point Likert scale (anchors: 0 = "never" and 4 = "almost always"). The PROMIS measures demonstrated good construct validity (intercept and slope equal or greater to 0.98) and internal consistency (pain interference, 4 items alpha = 0.85).
Brain imaging | This outcome will be measured at discharge from the program, which is approximately 3 weeks from the time of admittance.
  Structural and functional imaging will be acquired using resting-state functional magnetic resonance imaging (fMRI) scan. Motion will be censored using the Artifact Detection Tools (ART). Cortical masks derived from FreeSurfer will be used as seed regions for fMRI functional connectivity analysis. Time courses for the dorsolateral prefrontal cortex (DLPFC) will be extracted and used as a regressor to identify correlations with all other brain regions. Second-level analyses will be used to test differences in functional connectivity over time and between groups. All statistical tests will be corrected for multiple comparisons.
Functional disability | This outcome will be measured at discharge from the program, which is approximately 3 weeks from the time of admittance.
  The Functional Disability Inventory (FDI) will be administered to assess functional disability. Youth will rate their level of difficulty in completing daily activities in a variety of settings (e.g. home, school) on a 5-point Likert scale ranging from 0 "no trouble" to 4 "impossible." Higher scores are indicative of greater pain-related disability. The FDI has high internal consistency at baseline (alpha = .90) and post-treatment (alpha = .87).
Anxiety and Depressive Symptoms | This outcome will be measured at discharge from the program, which is approximately 3 weeks from the time of admittance.
  Anxiety and depressive symptoms will be assessed using the PROMIS Pediatric Profile-25 Anxiety and Depression subscales. Participants will report if they experienced any of the symptoms in the past 7 days using a 5-point Likert scale (anchors: 0 = "never" and 4 = "almost always"). The subscales have demonstrated good construct validity (intercept and slope equal to or greater than 0.93) and excellent internal consistency (depressive symptoms, 4 items, alpha = 0.91; anxiety symptoms, 4 items, alpha = 0.90).
Posttraumatic Stress Disorder (PTSD) Symptoms | This outcome will be measured at discharge from the program, which is approximately 3 weeks from the time of admittance.
  Youth PTSD symptomology will be assessed using the Child PTSD Symptom Scale (CPSS-V). The CPSS-V is a 20-item measure that maps on to the Diagnostic and Statistical Manual of Mental Disorders 5th Edition PTSD criteria, and assessed PTSD symptoms experienced by youth in the past month. Youth will be asked to identify something scary or upsetting that bothers them to think about. With that event in mind, they will be asked to respond to 20 items assessing PTSD symptoms on a 5-point Likert scale, ranging from "not at all" to "6 or more times a week/almost always." Total symptom severity scores are obtained by summing the 20 items (range: 0-80). A score of 31 or above indicates clinically elevated PTSD symptoms. The CPSS-V has excellent internal consistency, good test-retest reliability, and good convergent validity.
Pediatric Transcranial Magnetic Stimulation (TMS) Safety and Tolerability | This outcome will be measured at Day 6.
  Possible adverse events (headache, presyncope, nausea, etc.) will be screened and quantified as either mild, moderate, or severe. Any other potential side effects will be recorded and quantified.
Pediatric Transcranial Magnetic Stimulation (TMS) Safety and Tolerability | This outcome will be measured at Day 11.
  Possible adverse events (headache, presyncope, nausea, etc.) will be screened and quantified as either mild, moderate, or severe. Any other potential side effects will be recorded and quantified.

CONTACTS AND LOCATIONS:
Overall Officials: Jillian V Miller, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kashikar-Zuck S, Flowers SR, Claar RL, Guite JW, Logan DE, Lynch-Jordan AM, Palermo TM, Wilson AC. Clinical utility and validity of the Functional Disability Inventory among a multicenter sample of youth with chronic pain. Pain. 2011 Jul;152(7):1600-1607. doi: 10.1016/j.pain.2011.02.050. Epub 2011 Mar 31. PMID 21458162
- [Background] Noel M, Vinall J, Tomfohr-Madsen L, Holley AL, Wilson AC, Palermo TM. Sleep Mediates the Association Between PTSD Symptoms and Chronic Pain in Youth. J Pain. 2018 Jan;19(1):67-75. doi: 10.1016/j.jpain.2017.09.002. Epub 2017 Sep 27. PMID 28962895
- [Background] Vinall J, Pavlova M, Asmundson GJ, Rasic N, Noel M. Mental Health Comorbidities in Pediatric Chronic Pain: A Narrative Review of Epidemiology, Models, Neurobiological Mechanisms and Treatment. Children (Basel). 2016 Dec 2;3(4):40. doi: 10.3390/children3040040. PMID 27918444
- [Background] Perquin CW, Hazebroek-Kampschreur AAJM, Hunfeld JAM, Bohnen AM, van Suijlekom-Smit LWA, Passchier J, van der Wouden JC. Pain in children and adolescents: a common experience. Pain. 2000 Jul;87(1):51-58. doi: 10.1016/S0304-3959(00)00269-4. PMID 10863045
- [Background] Fearon P, Hotopf M. Relation between headache in childhood and physical and psychiatric symptoms in adulthood: national birth cohort study. BMJ. 2001 May 12;322(7295):1145. doi: 10.1136/bmj.322.7295.1145. PMID 11348907
- [Background] Shelby GD, Shirkey KC, Sherman AL, Beck JE, Haman K, Shears AR, Horst SN, Smith CA, Garber J, Walker LS. Functional abdominal pain in childhood and long-term vulnerability to anxiety disorders. Pediatrics. 2013 Sep;132(3):475-82. doi: 10.1542/peds.2012-2191. Epub 2013 Aug 12. PMID 23940244
- [Background] Hogan ME, Taddio A, Katz J, Shah V, Krahn M. Incremental health care costs for chronic pain in Ontario, Canada: a population-based matched cohort study of adolescents and adults using administrative data. Pain. 2016 Aug;157(8):1626-33. doi: 10.1097/j.pain.0000000000000561. PMID 26989805
- [Background] Eccleston C, Palermo TM, Williams AC, Lewandowski Holley A, Morley S, Fisher E, Law E. Psychological therapies for the management of chronic and recurrent pain in children and adolescents. Cochrane Database Syst Rev. 2014 May 5;2014(5):CD003968. doi: 10.1002/14651858.CD003968.pub4. PMID 24796681
- [Background] Hechler T, Kanstrup M, Holley AL, Simons LE, Wicksell R, Hirschfeld G, Zernikow B. Systematic Review on Intensive Interdisciplinary Pain Treatment of Children With Chronic Pain. Pediatrics. 2015 Jul;136(1):115-27. doi: 10.1542/peds.2014-3319. Epub 2015 Jun 22. PMID 26101358
- [Background] Hurtubise K, Blais S, Noel M, Brousselle A, Dallaire F, Rasic N, Camden C. Is It Worth It? A Comparison of an Intensive Interdisciplinary Pain Treatment and a Multimodal Treatment for Youths With Pain-related Disability. Clin J Pain. 2020 Nov;36(11):833-844. doi: 10.1097/AJP.0000000000000869. PMID 32769416
- [Background] Simons LE, Pielech M, Erpelding N, Linnman C, Moulton E, Sava S, Lebel A, Serrano P, Sethna N, Berde C, Becerra L, Borsook D. The responsive amygdala: treatment-induced alterations in functional connectivity in pediatric complex regional pain syndrome. Pain. 2014 Sep;155(9):1727-1742. doi: 10.1016/j.pain.2014.05.023. Epub 2014 May 23. PMID 24861582
- [Background] Glasser MF, Coalson TS, Robinson EC, Hacker CD, Harwell J, Yacoub E, Ugurbil K, Andersson J, Beckmann CF, Jenkinson M, Smith SM, Van Essen DC. A multi-modal parcellation of human cerebral cortex. Nature. 2016 Aug 11;536(7615):171-178. doi: 10.1038/nature18933. Epub 2016 Jul 20. PMID 27437579
- [Background] O'Reilly RC. The What and How of prefrontal cortical organization. Trends Neurosci. 2010 Aug;33(8):355-61. doi: 10.1016/j.tins.2010.05.002. Epub 2010 Jun 22. PMID 20573407
- [Background] Sallet J, Mars RB, Noonan MP, Neubert FX, Jbabdi S, O'Reilly JX, Filippini N, Thomas AG, Rushworth MF. The organization of dorsal frontal cortex in humans and macaques. J Neurosci. 2013 Jul 24;33(30):12255-74. doi: 10.1523/JNEUROSCI.5108-12.2013. PMID 23884933
- [Background] Bornhovd K, Quante M, Glauche V, Bromm B, Weiller C, Buchel C. Painful stimuli evoke different stimulus-response functions in the amygdala, prefrontal, insula and somatosensory cortex: a single-trial fMRI study. Brain. 2002 Jun;125(Pt 6):1326-36. doi: 10.1093/brain/awf137. PMID 12023321
- [Background] Seminowicz DA, Moayedi M. The Dorsolateral Prefrontal Cortex in Acute and Chronic Pain. J Pain. 2017 Sep;18(9):1027-1035. doi: 10.1016/j.jpain.2017.03.008. Epub 2017 Apr 8. PMID 28400293
- [Background] MacMaster FP, Croarkin PE, Wilkes TC, McLellan Q, Langevin LM, Jaworska N, Swansburg RM, Jasaui Y, Zewdie E, Ciechanski P, Kirton A. Repetitive Transcranial Magnetic Stimulation in Youth With Treatment Resistant Major Depression. Front Psychiatry. 2019 Mar 29;10:170. doi: 10.3389/fpsyt.2019.00170. eCollection 2019. PMID 30984044
- [Background] Zewdie E, Ciechanski P, Kuo HC, Giuffre A, Kahl C, King R, Cole L, Godfrey H, Seeger T, Swansburg R, Damji O, Rajapakse T, Hodge J, Nelson S, Selby B, Gan L, Jadavji Z, Larson JR, MacMaster F, Yang JF, Barlow K, Gorassini M, Brunton K, Kirton A. Safety and tolerability of transcranial magnetic and direct current stimulation in children: Prospective single center evidence from 3.5 million stimulations. Brain Stimul. 2020 May-Jun;13(3):565-575. doi: 10.1016/j.brs.2019.12.025. Epub 2019 Dec 30. PMID 32289678
- [Background] Fox MD, Liu H, Pascual-Leone A. Identification of reproducible individualized targets for treatment of depression with TMS based on intrinsic connectivity. Neuroimage. 2013 Feb 1;66:151-60. doi: 10.1016/j.neuroimage.2012.10.082. Epub 2012 Nov 7. PMID 23142067
- [Background] Garvey MA, Gilbert DL. Transcranial magnetic stimulation in children. Eur J Paediatr Neurol. 2004;8(1):7-19. doi: 10.1016/j.ejpn.2003.11.002. PMID 15023371